CLINICAL TRIAL: NCT00030537
Title: A Pilot Study to Evaluate Epidermal Growth Factor Receptor Signaling After Treatment With Oral OSI-774 in Patients With Locally Advanced or Metastatic Breast Cancer
Brief Title: Erlotinib in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069175; NCI-02-C-0061; NCI-5403; NCT00027313 (obsolete NCT alias)
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2002-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; stage IIIB breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor.

PURPOSE: Phase II trial to study the effectiveness of erlotinib in treating patients who have locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a change in epidermal growth factor receptor (EGFR) phosphorylation is detected in tumors of patients with locally advanced or metastatic breast cancer treated with erlotinib.
* Determine whether a change in other parameters of signal transduction that are downstream of EGFR (ERK and AKT) is detected in tumors of patients treated with this drug.
* Determine the toxicity of this drug in these patients.
* Determine the response duration and time to progression in patients treated with this drug.
* Correlate EGFR phosphorylation level with clinical findings and time to progression in patients treated with this drug.
* Correlate the pharmacokinetics of this drug with a change in EGFR phosphorylation in tumor biopsies of these patients.

OUTLINE: Patients receive oral erlotinib once daily. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed within 4 weeks.

PROJECTED ACCRUAL: A total of 15-20 patients will be accrued for this study within 7-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Locally advanced or metastatic disease
  * Incurable disease
* Tumor accessible for biopsy
* Prior breast cancer allowed
* No symptomatic or untreated brain metastases or carcinomatous meningitis

  * Neurologically stable patients with inactive brain metastases are allowed if off corticosteroids for at least 4 weeks prior to study
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* ALT/AST no greater than 2.5 times upper limit of normal

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* LVEF at least 40%
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Ophthalmic:

* No prior abnormalities of the cornea, including:

  * Dry eye syndrome or Sjogren's syndrome
  * Congenital abnormality (e.g., Fuch's dystrophy)
  * Abnormal slit-lamp examination with a vital dye (e.g., fluorescein or Bengal-Rose)
  * Abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* No concurrent use of contact lenses

Other:

* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to erlotinib (e.g., gefitinib or other anilinoquinazolines)
* No other concurrent uncontrolled illness
* No active infection
* No uncontrolled diabetes mellitus
* No psychiatric illness or social situation that would preclude study
* No untreated life-threatening disease
* No other primary malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* Weight less than 136 kg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 2 weeks since prior hormonal therapy
* No concurrent hormonal therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy except localized external beam radiotherapy for palliative treatment of metastatic disease (cannot include significant cardiac muscle within the radiotherapy field)

Surgery:

* Not specified

Other:

* No other concurrent investigational anticancer agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette R. Tan, MD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Center for Cancer Research, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland

REFERENCES:
- [Result] Tan AR, Yang X, Hewitt SM, Berman A, Lepper ER, Sparreboom A, Parr AL, Figg WD, Chow C, Steinberg SM, Bacharach SL, Whatley M, Carrasquillo JA, Brahim JS, Ettenberg SA, Lipkowitz S, Swain SM. Evaluation of biologic end points and pharmacokinetics in patients with metastatic breast cancer after treatment with erlotinib, an epidermal growth factor receptor tyrosine kinase inhibitor. J Clin Oncol. 2004 Aug 1;22(15):3080-90. doi: 10.1200/JCO.2004.08.189. PMID 15284258